CLINICAL TRIAL: NCT02313168
Title: F.R.O.N.T. Formula for Pre-operative Airway Assessment and Documentation
Status: Completed | Type: Observational
Sponsor: University of Debrecen (Other)
Collaborators: University of Zurich (Other); Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Tamas Vegh, MD, assistant professor anesthesiologist and intensive care specialist, University of Debrecen
Other Study IDs: AITT 2014/7; HBR/052/01763-2/2014 (Registry Identifier: Government Offices Public Health Administration Organization); DE KK RKEB/IKEB 4231-2014 (Other: Local Ethic Comittee University of Debrecen)
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2017-03

CONDITIONS: Difficult Airway
Keywords: difficult airway; prediction, FRONT score.
MeSH Terms: interventions — Observation; Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: preoperative FRONT score
  Interventions: Other: observation, inspection
- 2: intraoperative FRONT score
  Interventions: Other: observation, inspection

INTERVENTIONS:
Other: observation, inspection

SUMMARY:
The F.R.O.N.T. formula for pre-operative airway assessment and documentation

Background:

Prediction of difficult airway is one of the most important challenges before general anesthesia. Although in recent decades different scoring systems have been for the preoperative assessment of their sensitivity and specificity in predicting a difficult airway remains moderate. Recently, the calculation of composite scores using different formulae has been proposed as the most sensitive one. The aim of the present work was to test the clinical usefulness of the FRONT score, a recently developed scoring system.

Methods:

This study was a multi-center, inter-observer, prospective and double-blind investigation that included 976 patients from two university centers: 250 from the University of Cluj-Napoca, Romania, and 726 from the University of Debrecen, Hungary.

The preoperative evaluation of the patients was performed by a preoperative team of anesthesiologists (team A) who evaluated and scored the expected difficulty of the management of the airway. An intraoperative team of evaluators (team B) working independently from team A, performed the actual instrumentation of the airway and scored the actual findings. Both teams used the FRONT scoring system and worked independently from each other to ensure blinded assessment. Statistical analysis of the preoperative and intraoperative FRONT scores were performed post hoc.

DETAILED DESCRIPTION:
Criteria for preoperative assessment and grading for all five levels "F" 0 Normal level of difficulty or no difficulty to be expected

1. Difficulty to apply air tight the facial mask ventilation by one person (difficulty to maintain SpO2 above 92% with 100% O2), or inability to prevent the decrease in SpO2 during facial mask ventilation.
2. Increased ventilation difficulty, requiring the presence of two anesthetists in order to maintain the patient's oxygenation, or inability to ventilate the patient with the facial mask.

"R" 0 Normal level of difficulty or no difficulty to be expected

1. Incomplete teeth, loose teeth, edentulous status, incisor protrusion, prognathia, micrognathia, limited opening of the mouth but still more than 3 cm., expected difficulty with direct laringoscopy and/or insertion of a supraglottic device.
2. Mobile teeth, mouth opening less than 3 cm, laryngoscopy or insertion of a supraglottic airway device impossible "O"

0 Normal level of difficulty or no difficulty to be expected

1 Laryngoscopy and intubation difficult expected by intaroral mass, abscess, anatomical anomalies (large tongue) 2 Laryngoscopy and tracheal intubation expected to be extremely difficult or impossible "N" 0 Normal level of difficulty or no difficulty to be expected

1. Reduced mobility of the cervical spine, short neck, bulky chest, special positioning of the patient necessary (roll under the shoulders)
2. Immobile cervical spine "T"

0 Normal level of difficulty or no difficulty to be expected

1. Expected trouble for passing the tube through the glottis (polyp, tumor, abscess), and tube with smaller diameter necessary
2. Severe obstruction in the upper airway (polyp, tumor, abscess, paralysis of the vocal cords), tracheal stenosis, tracheomalacia

Criteria for intraoperative assessment and grading for all five levels. "F" 0 Normal level of difficulty or no difficulty

1. Difficulty to seal the face mask accordingly by one person in order to maintain SpO2 above 92% by ventilating with oxygen.
2. Inability to maintain SpO2 above 92% by ventilating with oxygen with handling the face mask by two persons.

"R" 0 Normal level of difficulty or no difficulty

1. Incomplete dentition, protruding incisives, prognathia, micrognathia, a reduced interincisive gap above 3 cm thus explicitly hampering (but not completely preventing) intubation or supraglottic device insertion.
2. Incomplete dentition, protruding incisives, prognathia, micrognathia, a reduced interincisive gap below 3 cm limiting intubation or supraglottic device insertion.

"O" 0 Normal level of difficulty or no difficulty

1. Macroglossia, presence of tumours or other findings with increased oral tissue mass, tongue base processes which hamper the performance of direct laryngoscopy (Cormack/Lehane grades up to 3°), conventional intubation or the insertion of a supraglottic airway. Final success could be achieved after two attempts to secure the airway with any adopted technique.
2. Macroglossia, presence of tumours or other findings with increased oral tissue mass, tongue base processes which prevent the performance of direct laryngoscopy (Cormack/Lehane grade 4°), conventional intubation or the insertion of a supraglottic airway. Tracheal intubation could be achieved only after recurring to a visualizing technique (e.g. flexible fiberoptic).

"N" 0 Normal level of difficulty or no difficulty

1. Reduced cervical spine mobility, short neck, risk of spinal cord damage by certain head positions that hamper direct laryngoscopy and conventional means of tracheal intubation. Successful intubation possible by 2 or more attempts. Supraglottic airway insertion is not affected.
2. Reduced cervical spine mobility, short neck, risk of spinal cord damage by certain head positions that prevent direct laryngoscopy and conventional means of tracheal intubation. Tracheal intubation could be achieved only after recurring to a visualizing technique (e.g. flexible fiberoptic). Supraglottic airway insertion may have been affected.

"T" 0 Normal level of difficulty or no difficulty

1. Difficult forwarding of a tracheal tube with regular diameter to a mid-tracheal position. Supraglottic airway insertion is not affected.
2. Impossible forwarding of a tracheal tube even with a reduced diameter to a mid-tracheal position. Supraglottic airway insertion is not affected but ventilation is difficult or impossible. Necessity to apply jet ventilation or to bypass the oro-tracheal route by performing a trans-tracheal access.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older going to be intubated for general anesthesia for elective operation

Exclusion Criteria:

age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients (over 18 years) going elective surgery.
Sampling Method: Probability Sample
Enrollment: 1150 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Correlation between the preoperative and the intraoperative FRONT scores. | 2 weeks (between the preop. anesthesiological examination and the operation)
  The preoperative evaluation of the patients was performed by a preoperative team of anesthesiologists (team A) who evaluated and scored the expected difficulty of the management of the airway. An intraoperative team of evaluators (team B) working independently from team A, performed the actual instrumentation of the airway and scored the actual findings. Both teams used the FRONT scoring system and worked independently from each other to ensure blinded assessment. Statistical analysis of the preoperative and intraoperative FRONT scores will be performed post hoc. (correlation analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Bél Mr Fülesdi, MD, PhD, DSci, Principal Investigator — Hungary University of Debrecen Debrecen, Hungary, 4032
Locations (1):
- Hungary University of Debrecen, Debrecen, Hajdú-Bihar, Hungary